CLINICAL TRIAL: NCT06462742
Title: Microwave Ablation Versus Liver Resection for Intrahepatic Cholangiocarcinoma Within Milan Criteria
Brief Title: Microwave Ablation Versus Liver Resection for Intrahepatic Cholangiocarcinoma
Acronym: MALRIC
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Other Study IDs: S2024-0606
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Overall Survival; Disease-free Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MWA: iCCA patients who underwent microwave ablation (MWA).
  Interventions: Procedure: Microwave ablation (MWA) versus Liver Resection (LR)
- LR: iCCA patients who underwent liver resection (LR)
  Interventions: Procedure: Microwave ablation (MWA) versus Liver Resection (LR)

INTERVENTIONS:
Procedure: Microwave ablation (MWA) versus Liver Resection (LR) — Microwave ablation (MWA) is one of the newer modality of thermal ablation and has proven its safety and efficacy in the management of the tumors amenable for ablation for primary and metastatic diseases.
  Liver resection is a surgery to remove part of the liver to eradicate tumors.

SUMMARY:
Thermal ablation has been recommended by worldwide guidelines as first-line treatment for hepatocellular carcinoma (HCC), while evidence regarding its efficacy for primary intrahepatic cholangiocarcinoma (iCCA) is lacking. The goal of this observational study is to study the efficacy of ablation in treating iCCA by comparing its prognosis with surgery. The main questions it aims to answer are:

* Whether microwave ablation could achieve similar efficacy with liver resection in treating iCCA
* What is the risk factor for ablation or surgery in treating iCCA
* What kind of iCCA patients could receive ablation as their first-line treatment In this real-world multicenter cohort study, we will collect data of iCCA patients from hospitals who underwent microwave ablation (MWA) or liver resection (LR) for tumors within Milan criteria. Survival will be compared between patients treated by MWA or LR.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically diagnosed iCCA based on the WHO classifications;
2. curative-intent liver resection or microwave ablation;
3. tumor within Milan criteria, namely single tumor ≤5cm in maximum diameter; multiple tumors ≤3 in number and each ≤3cm; no evidence of major vascular/hilar invasion, extrahepatic/lymphatic metastasis or other malignancies;
4. age ≥18 years.

Exclusion Criteria:

Patients not meeting any one of the inclusion criteria were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients pathologically diagnosed with intrahepatic cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | More than 3 years]
  OS was defined as death related to any cause and was indexed from the date of ablation or surgery until last contact or death
Disease-free survival | More than 3 years
  DFS was defined as the time interval between first treatment and recurrence or death, whichever occurred earlier.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No